CLINICAL TRIAL: NCT01192256
Title: Does Smoking Status After Being Diagnosed With Lung Cancer Influence Outcome? An Observational Cohort Study.
Brief Title: Studies Examining the Importance of Smoking After Being Diagnosed With Lung Cancer
Acronym: LungCast
Status: Completed | Type: Observational
Sponsor: Dr Keir Lewis (Other)
Collaborators: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor-Investigator, Dr Keir Lewis, Professor in Medicine and Consultant Chest Physician, Hywel Dda Health Board
Organization: Hywel Dda Health Board (Other)
Other Study IDs: 09/WMW01/28; WS763986 (Other Grant/Funding Number: GRAND Pfizer)
Record Dates: First submitted 2010-08-27; First posted 2010-09-01 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Lung Cancer
Keywords: smoking; cessation; mortality; quality of life
MeSH Terms: conditions — Lung Neoplasms; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A large project consisting of:

a) an observational trial where smoking status is recorded on 1400 consecutive people newly diagnosed with lung cancer. Smoking status is biologically validated with exhaled carbon monoxide (eCO) levels every 3 months. Survival, cancer progression and treatment complications will be recorded and compared in smokers, ex-smokers and never smokers.

DETAILED DESCRIPTION:
Smoking causes around 85% of lung cancer. Continued smoking after diagnosis probably worsens survival and increases treatment complications but prospective well-designed studies are lacking.

This project is an observational cohort study recording outcomes in smokers, never-smokers, and ex-smokers, using exhaled carbon monoxide to validate smoking status when they attend for further lung cancer clinics.

This project is unique, as every patient with a clinical diagnosis of lung cancer will have their smoking status biologically validated by a quick and easy test, and those enrolled in the smoking cessation treatments or not will also complete a generic quality of life questionnaire at regular intervals. These appointments will coincide with other hospital appointments wherever possible, and survival status will reported up to 24 months after enrolment.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of lung cancer

Exclusion Criteria:

* refusal Consent
* inability to provide exhaled CO
* active psychiatric illness or substance misuse
* concurrent malignancies of another type other than non-melanoma skin cancer
* unable to travel for sessions with smoking cessation counsellor and / or outpatient visits from outset
* WHO performance status 4
* Life expectancy less than 6 weeks.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Median and 2-year survival rates in confirmed smokers versus non- smokers newly diagnosed with lung cancer. | 24 months

SECONDARY OUTCOMES:
Median survival and 2-year survival rates by smoking status for early (Stage I/II NSCLC) versus those with advanced (Stage III/IV) NSCLC. | 24 months
Number of treatment complications in smokers versus non-smokers (frequency surgical wound complications, radiotherapy induced pneumonitis and median total radiation (Gy) dose; frequency and duration of neutropenic sepses | 2 years
Point prevalence of smoking at 0, 3, 6 12, 24 months | 2 years
Comparison of changes in health related quality of life (EQ5D) in smokers versus non-smokers | 2 years
Accrual and attendance rates of lung cancer patients attending a hospital smoking cessation service | 2 years
Estimate of cost per quality adjusted life year gained by smoking cessation advice in both quit strategies for smokers | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Keir E Lewis, MD, Principal Investigator — Hywel Dda
Locations (2):
- United Kingdom (2):
  - Llandough Hospital, Cardiff and Vale University Health Board, Cardiff, Wales
  - Hywel Dda Health Board, Llanelli, Wales

REFERENCES:
- [Result] Gemine RE, Ghosal R, Collier G, Parry D, Campbell I, Davies G, Davies K, Lewis KE; LungCast Investigators. Longitudinal study to assess impact of smoking at diagnosis and quitting on 1-year survival for people with non-small cell lung cancer. Lung Cancer. 2019 Mar;129:1-7. doi: 10.1016/j.lungcan.2018.12.028. Epub 2018 Dec 28. PMID 30797485
- [Derived] Gemine RE, Davies GR, Lanyon K, Rees SE, Campbell I, Lewis KE; LungCAST Investigators. Quitting smoking improves two-year survival after a diagnosis of non-small cell lung cancer. Lung Cancer. 2023 Dec;186:107388. doi: 10.1016/j.lungcan.2023.107388. Epub 2023 Oct 1. PMID 37820539
- [Derived] Jones M, Lowin J, Sewell B, Gemine RE, Rees SE, Lanyon K, Lewis KE. The Economic Potential of Smoking Cessation Interventions at the Point of Diagnosis of Non-Small Cell Lung Cancer. Value Health. 2023 Aug;26(8):1192-1200. doi: 10.1016/j.jval.2023.03.2429. Epub 2023 Apr 12. PMID 37059391